CLINICAL TRIAL: NCT00006082
Title: Open Label Phase II Study on RFS 2000 (9-Nitro-Camptothecin, 9-NC) Administered as a "5 Days On - 2 Days Off" Oral Treatment in Advanced Small Cell Lung Cancer
Brief Title: Nitrocamptothecin in Treating Patients With Advanced Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16996SL; EORTC-16996SL
Record Dates: First submitted 2000-08-03; First posted 2003-05-22 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — rubitecan

INTERVENTIONS:
Drug: rubitecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of nitrocamptothecin in treating patients who have advanced small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response and duration of objective response in patients with advanced small cell lung cancer treated with nitrocamptothecin.
* Determine the probability of objective response as expressed by the response rate in patients treated with this regimen.
* Determine the toxicities of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to disease status (sensitive vs refractory).

Patients receive oral nitrocamptothecin daily for 5 consecutive days each week for 3 weeks. Treatment continues every 3 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve stable disease (SD) receive up to 4 additional courses past SD. Patients who achieve partial response (PR) or complete response (CR) receive a minimum of 2 additional courses past CR or PR.

Patients are followed every 6 weeks until disease progression or initiation of another antitumor treatment.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for the sensitive disease stratum and a total of 19-24 patients will be accrued for the refractory disease stratum

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven advanced (extensive stage) small cell lung cancer with progressive or recurrent disease after 1 first line chemotherapy regimen

  * Sensitive disease, defined as a response to prior chemotherapy lasting at least 3 months from the end of all prior treatment, including radiotherapy, until the time of progression OR
  * Refractory disease, defined as no response to prior chemotherapy, or a response to prior chemotherapy followed by progression within 3 months after completion of all prior therapy, including radiotherapy
* Minimum of 1 target lesion that can be accurately measured in at least 1 dimension

  * 20 mm or more with conventional techniques OR
  * 10 mm or more with spiral CT scans
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase, SGOT, and SGPT no greater than 2.5 time ULN (no greater than 5 times ULN if hepatic metastases present)

Renal:

* Creatinine no greater than 1.7 mg/dL

Cardiovascular:

* No ischemic heart disease within the past 6 months
* Normal 12 lead electrocardiogram

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior or concurrent malignancy except cone biopsied carcinoma of the cervix or adequately treated basal cell or squamous cell skin cancer
* No unstable systemic disease or active uncontrolled infection
* No psychological, familial, sociological, or geographical condition that may preclude compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior maintenance therapy with biologic agents following first line chemotherapy allowed
* No concurrent filgrastim (G-CSF) with nitrocamptothecin

Chemotherapy:

* See Disease Characteristics
* Greater than 4 weeks since prior chemotherapy
* No more than 1 prior chemotherapy regimen for extensive disease
* Alternate or sequential use of different regimens without interruption in first line treatment is considered 1 first line therapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* Greater than 4 weeks since prior radiotherapy

Surgery:

* Greater than 2 weeks since prior major surgery

Other:

* No other concurrent anticancer therapy
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2000-05; Primary Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fumoleau, MD, PhD, Study Chair — Centre Georges Francois Leclerc
Locations (1):
- CRLCC Nantes - Atlantique, Nantes-Saint Herblain, France